CLINICAL TRIAL: NCT02298439
Title: Non-Alcoholic Fatty Liver Disease Patient Registry
Brief Title: Fatty Liver Patient Registry
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Johane Allard, MD, FRCPC, University Health Network, Toronto
Other Study IDs: 13-6128-AE
Record Dates: First submitted 2014-10-24; First posted 2014-11-24 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the Non-Alcoholic Fatty Liver Disease (NAFLD) registry is to collect demographic and clinical data on patients being treated for NAFLD and to determine the factors affecting the progression of the disease as well as the success of different treatment strategies.

DETAILED DESCRIPTION:
The NAFLD registry is a local database provided by the principal investigator, Dr. J. Allard, which will be stored on the Research Intranet at the University Health Network, Toronto. The database will be password protected. Only clinic personnel and members of Dr. Allard's research team involved in the study will have access to the database. A code and date of birth will be used to identify each patient. All patients entering the NAFLD clinic at Toronto General Hospital will be consented for the registry. Only data from their regular clinic visits will be used for entry into the registry. Data entered into the registry will include: 1) Patient demography: age, sex, ethnicity, medical history; 2) Anthropometry: weight, height, BMI, waist circumference; 3) Nutritional assessment: Food records and food frequency questionnaires are kept by the subjects and data will be analyzed to assess the intake of macro- and micronutrients. Amount of alcohol and number of cigarette smoked will also be recorded; 4) Physical Activity will be assessed using the Paffenbarger Physical Activity Questionnaire; 5) Medications: insulin, non-steroidal anti-inflammatory drugs, corticosteroids, statins, medications used to treat diabetes/obesity (e.g. metformin, thiazolidinediones, orlistat…), medication to treat liver disease (eg. urso, carnitine, choline…), antioxidant vitamin or fish oil supplementation; 6) Blood work, currently including: complete blood count, biochemistry including liver enzymes, total protein, albumin, glucose, insulin, and blood lipid profile; other diagnostic blood work done to exclude other causes of liver disease, e.g. ceruloplasmin, anti-smooth muscle antibodies,… One plasma sample will be stored for assessment of cytokeratin 18 (CK-18) fragments as a novel marker for NASH in patients with NAFLD; 7) Presence of metabolic syndrome; 8) Disease categorization: SS, NASH, cirrhosis; 9) Survival: alive, death: causes, NAFLD-related or not NAFLD-related; 10) Liver biopsy results, NAFLD fibrosis score, and elastography results.

Data will be entered after every clinic visit. Case report forms will be used to collect the data from the patient charts and facilitate data input into the registry database All patients will be followed prospectively until withdrawal from the clinic or death. Descriptive statistics will be performed. For the entire NAFLD population, probability of survival, cirrhosis, as well as liver and non-liver related morbidity will be calculated using the Kaplan Meier method.

ELIGIBILITY:
Inclusion Criteria:

- Patients being treated for NAFLD at the Toronto General Hospital NAFLD clinic

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Non-Alcoholic Fatty Liver Disease (NAFLD )which includes simple steatosis (SS) and non-alcoholic steatohepatitis (NASH) that being treated
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Disease categorization | Baseline
  Specific diagnosis of NAFLD: simple steatosis (SS), steatohepatitis (NASH), cirrhosis

SECONDARY OUTCOMES:
Disease categorization | at each clinic visit, up to 5 years
  Specific diagnosis of NAFLD: simple steatosis (SS), steatohepatitis (NASH), cirrhosis
Liver biopsy results | at each clinic visit, up to 5 years
  NAFLD fibrosis score, and elastography results
Survival | at each clinic visit, up to 5 years
  Alive, death: causes, NAFLD-related or not

OTHER OUTCOMES:
Patient demography | at each clinic visit, up to 5 years
  Age, sex, ethnicity, medical history from medical chart
Anthropometry | at each clinic visit, up to 5 years
  Body mass index, waist circumference
Macro- and micronutrient intake | at each clinic visit, up to 5 years
  Food records and food frequency questionnaires
Physical activity | at each clinic visit, up to 5 years
  Paffenbarger Physical Activity Questionnaire
Presence of metabolic syndrome | at each clinic visit, up to 5 years
Medications | at each clinic visit, up to 5 years
  From clinical chart
Complete Blood Cell Count | at each clinic visit, up to 5 years
  Routine laboratory test
Biochemistry | at each clinic visit, up to 5 years
  Liver enzymes, total protein, albumin, glucose, insulin, and blood lipid
NAFLD specific diagnostic blood work | at each clinic visit, up to 5 years
  Ceruloplasmin, anti-smooth muscle antibodies
Cytokeratin 18 | at each clinic visit, up to 5 years
  CK-18 fragments

CONTACTS AND LOCATIONS:
Overall Officials: Johane Allard, MD, FRCPC, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Schwenger KJ, Allard JP. Clinical approaches to non-alcoholic fatty liver disease. World J Gastroenterol. 2014 Feb 21;20(7):1712-23. doi: 10.3748/wjg.v20.i7.1712. PMID 24587650
- [Result] Monteiro J, Leslie M, Moghadasian MH, Arendt BM, Allard JP, Ma DW. The role of n - 6 and n - 3 polyunsaturated fatty acids in the manifestation of the metabolic syndrome in cardiovascular disease and non-alcoholic fatty liver disease. Food Funct. 2014 Mar;5(3):426-35. doi: 10.1039/c3fo60551e. PMID 24496399
- [Result] Allard JP, Aghdassi E, Mohammed S, Raman M, Avand G, Arendt BM, Jalali P, Kandasamy T, Prayitno N, Sherman M, Guindi M, Ma DW, Heathcote JE. Nutritional assessment and hepatic fatty acid composition in non-alcoholic fatty liver disease (NAFLD): a cross-sectional study. J Hepatol. 2008 Feb;48(2):300-7. doi: 10.1016/j.jhep.2007.09.009. Epub 2007 Nov 20. PMID 18086506
- [Result] Raman M, Allard J. Non alcoholic fatty liver disease: a clinical approach and review. Can J Gastroenterol. 2006 May;20(5):345-9. doi: 10.1155/2006/918262. PMID 16691301
- [Result] Allard JP. Other disease associations with non-alcoholic fatty liver disease (NAFLD). Best Pract Res Clin Gastroenterol. 2002 Oct;16(5):783-95. doi: 10.1053/bega.2002.0330. PMID 12406445